CLINICAL TRIAL: NCT06956313
Title: Hydraulic Pressure Sinus Lift Versus Piezoelectric Lift Via Lateral Approach: A Randomized Controlled Clinical Trial.
Brief Title: Hydraulic Pressure Lateral Sinus Lift Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPLT-4-25
Record Dates: First submitted 2025-05-01; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Sinus Lifting; Piezoelectric Technique
Keywords: advanced intelligence drill; Sinus lift; hydraulic pressure sinus lift; external sinus lift,; piezoelectric surgery; lateral approach

STUDY DESIGN:
Who Masked: Investigator
Masking Description: patients were allocated in a 1:1 ratio using an on-site computer software system with concealed allocation through sequentially numbered, opaque, sealed envelopes (SNOSE). This was a double-blind study, so neither the statistical analyst nor the patients were aware of the surgical procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPLT Group (Experimental): patients with posterior deficient maxilla managed with osteotomy for lateral sinus floor augmentation using the Hydraulic Pressure Lifting Technique with A.I drill and hydraulic-powered Aqua-Lifter (OLA system) were assigned to HPLT Group
  Interventions: Device: Hydraulic Pressure Lifting Technique
- PSLT Group (Experimental): posterior deficient maxilla managed with osteotomy for lateral sinus floor augmentation using Piezo-Surgical Lifting Technique were assigned to PSLT Group
  Interventions: Device: Piezo-Surgical Lifting Technique

INTERVENTIONS:
Device: Hydraulic Pressure Lifting Technique — Hydraulic Pressure Lifting Technique
  Arms: HPLT Group
Device: Piezo-Surgical Lifting Technique — Piezo-Surgical Lifting Technique
  Arms: PSLT Group

SUMMARY:
the study aims to assess the effectiveness of hydraulic pressure sinus lift via lateral wall approach, versus piezoelectric surgery in patients with deficient posterior maxilla.

DETAILED DESCRIPTION:
This study involves a randomized clinical trial of 20 participants with less than 6 mm bone height in the posterior maxilla in need of Maxillary Sinus Floor Augmentation using the lateral window approach. Patients will be randomly assigned to two groups; the HPLT Group which include 10 patients who will undergo hydraulic pressure for osteotomy preparation for lateral sinus lifting technique, and the PSLT Group which include 10 patients managed using piezoelectric surgery. Clinical and radiographic assessment of bone augmentation, as well as intraoperative biological complications and postoperative complications were recorded.

ELIGIBILITY:
Inclusion Criteria:

* The study included patient with deficient posterior maxilla with less than 6mm of bone height conﬁrmed by a pre-operative tomographic scan. All healthy (ASA I, II) non- smoker patients were eligible for the study. The absence of uncontrolled diabetes, systemic illnesses, sinusitis, immune deficiency disorders, were also required for inclusion.

Exclusion Criteria:

* Patients with sinus infection, neoplasm or a large cyst of the sinus, or those who previously underwent a Caldwell-Luc surgery for the same surgical site were excluded

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
radiographic appraisal of gain in alveolar bone height | 6 months
  Postoperative radiographic appraisal was conducted by an immediate postoperative CBCT, followed by other one after 6 postoperative month's. Measurements of the bone height was conducted from the alveolar crest to the floor of the maxillary sinus on a cross-section view of the CBCT (Carestream Health, Rochester, NY). Radiographic assessment of the amount of bone height gain in 6 months period was performed by comparing the bone height measurements between the 6 postoperative months' CBCT with the preoperative scan.

SECONDARY OUTCOMES:
incidence of membrane perforation | Until the end of the operation
  incidence of membrane perforation during the operation was assessed in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study
Supporting Information: SAP